CLINICAL TRIAL: NCT02521675
Title: Multicentre Randomized Cross-over Study Assessing in Type 1 Diabetic Patients With Pump Insulin the Non-inferiority of Glycemic Control Obtained With the Algorithms Tested in DIABRASPORT Versus the Rest Period Without Physical Activity
Brief Title: Validation of Algorithms for Basal Insulin Rate Reductions in Type 1 Diabetic Patients Practising Physical Activity in Real Life Conditions
Acronym: Diabrasport2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-A00709-40
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type I; Adjustment of Basal Insulin Flow Rate During Physical Activity; Adjustment of Prandial Insulin in Case of Physical Activity
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabrasport then Rest (Other): Between each period, the patient should respect a wash-out period of at least one week, during which they will be asked not to practice physical activity.
  Interventions: Behavioral: Usual algorithm; Behavioral: Diabrasport algorithm; Behavioral: Rest; Device: Holter Glycemic Ipro2, Medtronic
- Rest then Diabrasport (Other): Between each period, the patient should respect a wash-out period of at least one week, during which they will be asked not to practice physical activity.
  Interventions: Behavioral: Usual algorithm; Behavioral: Diabrasport algorithm; Behavioral: Rest; Device: Holter Glycemic Ipro2, Medtronic

INTERVENTIONS:
Behavioral: Usual algorithm — The patient will be fitted with a CGMS (continuous glucose monitoring system) (data not shown) and it will be given the booklet to collect events + food survey
  The patient goes home and he must perform 3 physical activities during the week (30-60 minutes) using its usual algorithms (glucose administration or adaptation of the BR), in the afternoon, and spacing them at least 24 hours :
  * Moderate activity 3 hours after lunch
  * Intense activity 3 hours after lunch
  * Moderate activity 90 min after lunch These activities should not exceed 1 hour in wherever possible
Behavioral: Diabrasport algorithm — The patient will be fitted with a CGMS (data not shown) and it will be given the booklet to collect events + food survey
  The patient goes home and he must perform 3 physical activities during the week (identical to those carried out during the week "test algorithms usual" and during comparable periods) using DIABRASPORT algorithms, the afternoon and in the spacing at least 24 hours:
  * Moderate activity 3 hours after lunch
  * Intense activity 3 hours after lunch
  * Moderate activity 90min after lunch These activities shall not exceed one hour
Behavioral: Rest — The patient will be fitted with a CGMS (data not shown) and it will be given the booklet to collect events + food survey.
  The patient goes home and he will not perform any physical activity during the week
Device: Holter Glycemic Ipro2, Medtronic

SUMMARY:
There is no specific recommendations on the adjustments of the insulin treatment in the event of physical activity (PA) in T1D patients treated on insulin pump therapy. Patients often prefer additional carbohydrates intake rather than the reduction of their insulin doses because of the lack of specific algorithms.

The DIABRASPORT 2 study aims to demonstrate that using algorithms DIABRASPORT, during a week of physical activity (PA), the incidence of hypoglycaemia is not different from that obtained during a week of rest without physical activity.

It is a multi-center European, controlled, randomized, cross-over, study, in 100 T1D patients practicing an occasional AP.

25 centers involved in this study.

After agreeing to participate in the study, patients will read the information leaflet, ask questions to the investigator physician and they will date and sign the consent form. The investigator physician will do the same.

They will be then drawn randomly via the electronic CRF (eCRF) to determine the order in which they will realize the rest vs DIABRASPORT sessions.

The study will take place in 5 weeks:

During the weeks Baseline and Diabrasport, patients will have to make 3 physical activity of 30 to 60 minutes separated by at least 24 hours:

* moderate activity 3 hours after lunch
* intense activity 3 hours after lunch
* activity moderate 90 min after lunch They will use their usual algorithms (Cho intake or adjustment of the dose of insulin) during the week Baseline and they will use the Diabrasport algorithm during the week Diabrasport.

Patients will be equipped with a holter Glycemic iPro2, Medtronic, whose data are hidden.

During the week of rest, patients should do no physical activity during the week. They will be equipped with the Glycemic holter.

Patients will have to fill a food survey the days they practice PA. Between each period, the patient must respect a period of wash-out for one week at least, during which he will be asked to not practice physical activity.

Validation of algorithms simple, easy to implement, adaptable by patients, could help to improve balance metabolic and practice of sport among the T1D.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years
* Patient with type 1 diabetes for at least 1 year
* Patient receiving insulin pump under basal-prandial regimen for at least 3 months
* Patient practicing functional insulin therapy, or using a fixed plane defined food
* Patients with a stable basal rate for at least 1 week
* Patient practicing regular physical activity and reproducible identically
* Patient with HbA1c older than 3 months between 6.5% and 9.5% (HbA1c ≤ 6.5% ≤ 9.5%)
* Patients with BMI ≤ 35
* Patient who agreed to participate in the study and who signed an informed consent
* Patient not participating in another protocol
* Patient covered by social security

Exclusion Criteria:

* Patients with a history of severe hypoglycemia without accidental cause in the 6 months preceding the entry in the protocol
* Patient not receiving its hypoglycaemia below the threshold of 0.5 g / L
* Patient with perforating foot ulcer or a known history of heart disease or obliterative arteriopathy of the lower limbs, or a history of cerebrovascular accident, or ongoing proliferative retinopathy or renal failure
* Patient with poorly controlled hypertension
* Pregnant woman
* Patients deprived of liberty by judicial or administrative decision, patients placed under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
the number of hypoglycemic events, defined by any threshold crossing 60 mg / dL (3.33mmol / L), measured in the interstitial glucose sensor continuously over a period of 24h | 24h
percentage of time spent over 24 hours in the euglycemic range [70; 180] mg / dL ([3.89, 10] mmol / L) | 24h
percentage of time spent over 24 hours in hyperglycemia (> 180 mg / dL) (> 10 mmol / L) | 24h

SECONDARY OUTCOMES:
Number of hypoglycemic events, defined by any threshold crossing 70 mg / dL (3.9 mml / L), and <54 mg / dL (3 mmol / l) measured by interstitial continuous glucose sensors | 1 week
Number of hyperglycemic events, defined by any crossing of the threshold of 180 mg / dL (10 mml / L), measured by continuous interstitial glucose sensors. | 1 week
Metabolic goals analysis: | 1 week
  * percentage of time spent in the intervals [70; 180] and [80; 140] mg / dL, [3.89; 10] and [4.44; 7.78] mmol / L
  * percentage of time passes hypoglycemia (<60mg / dL) (<3.33 mmol / L)
  * percentage of time spent in hypoglycemia (<54mg / dL) (<3 mmol / L)
  * percentage of time spent in hypoglycemia (<70mg / dL) (<3.89 mmol / L)
  * percentage of time spent <80 mg / dL; (<4.44 mmol / L)
  * percentage of time spent in hyperglycemia (> 180 mg / dL) (> 10 mmol / L)
  * percentage of time spent> 140 mg / dL (> 7.78 mmol / L)
Nadirs analysis of blood glucose during the night (value reached) | 1 week
Nadirs analysis of blood glucose during the night (time to onset) | 1 week
Analysis of quantities of glucose administration consumed during and at the waning of physical activity | 1 week
Comparison of average values of continuous glucose measurements according to the period (DIABRASPORT, rest and Baseline) and at different times of the day and night. | 1 week
Analysis by subgroups, depending on the type of physical activity and its duration, a link between a typology of physical activity or patients, and the number of hypoglycemia events during or waning of physical activity | 1 week
Analysis of evaluation questionnaires intensity PA (Borg) and quality of life (EVA) | 1 week
Comparison between number of hypoglycemic events predicted by the prediction function "DIABRASPORT" and number of hypoglycemic events actually occurred. | 1 week

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Hôpital Universitaire, Angers
  - Hôpital Henri Duffaut, Avignon
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Universitaire, Brest
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - Centre Hospitalier Louis Pasteur, Dole
  - Centre Hospitalier, Douai
  - Hôpital Universitaire, Grenoble
  - Fondation Hôtel Dieu du Creusot, Le Creusot
  - Centre Hospitalier Régional Universitaire, Lille
  - Centre Hospitalier Universitaire, Lyon
  - Hôpital de la Conception, Marseille
  - Mérignac
  - Centre Hospitalier Universitaire, Rennes
  - Centre Hospitalier, Saint-Dié
  - Centre Hospitalier Régional Universitaire, Strasbourg
  - Hôpital Jean Bernard, Valenciennes